CLINICAL TRIAL: NCT04364204
Title: Hypothermia Prevention in Low Birthweight and Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of South Carolina (Other)
Collaborators: Centre for Learning and Childhood Development - Ghana (Unknown); Ghana Health Services (Other Government); Korle-Bu Teaching Hospital, Accra, Ghana (Other)
Responsible Party: Principal Investigator, Mufaro Kanyangarara, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00095600
Record Dates: First submitted 2020-03-16; First posted 2020-04-28 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Neonatal Hypothermia
Keywords: newborn; low birthweight; kangaroo mother care
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo mother care with bracelet (Experimental)
  Interventions: Other: Kangaroo Mother Care and BEMPU bracelet
- Kangaroo mother care (Active Comparator)
  Interventions: Other: Kangaroo Mother Care

INTERVENTIONS:
Other: Kangaroo Mother Care and BEMPU bracelet — Kangaroo mother care involves early, continuous and prolonged skin-to-skin contact between a mother and her newborn, frequent and exclusive breastfeeding and early discharge from hospital. The BEMPU bracelet, also known as the BEMPU Tempwatch, is a silicone band with a thermistor metal cup that emits an audio alarm and flashes an orange light when the body temperature drops below 36.5⁰C, signaling hypothermia and prompting caregiver to provide thermal care.
  Arms: Kangaroo mother care with bracelet
Other: Kangaroo Mother Care — Kangaroo mother care involves early, continuous and prolonged skin-to-skin contact between a mother and her newborn, frequent and exclusive breastfeeding and early discharge from hospital. This is the current standard of care for low birthweight/preterm infants.
  Arms: Kangaroo mother care

SUMMARY:
Preterm birth complications are the leading cause of neonatal mortality and account for over one million neonatal deaths annually. About 12% of babies are born before 37 weeks of gestation, and are at risk for hypothermia, hypoglycemia, infections, and mortality during the first 28 days of life. Kangaroo Mother Care (KMC) has been shown to reduce hypothermia, neonatal infections and neonatal mortality, while improving weight gain and mother-infant attachment; however, implementation to scale has been slow. The BEMPU® bracelet offers the opportunity to monitor the body temperature of newborns for the early detection of hypothermia and to increase the uptake of KMC. Further research is needed to evaluate the impact of the BEMPU® bracelet on KMC practices and neonatal health outcomes and facilitate its adoption in low-resource settings. The goal of this research is to evaluate its effect on KMC practices and neonatal health outcomes in Ghana. Evidence of a significant impact on outcomes will provide critical evidence to facilitate prompt identification of hypothermia, maximize the benefits of KMC, decrease the risk of neonatal death, and impact the leading cause of neonatal mortality in Ghana and other settings.

DETAILED DESCRIPTION:
This study will evaluate the effect of the bracelet on KMC practices and neonatal health outcomes in LBW infants using a randomized controlled trial. Infants currently being treated in the KMC or neonatal wards of the participating hospitals will be screened for eligibility by study nurses. After obtaining parental consent, infants will be randomly assigned with a 1:1 ratio to KMC with and without the BEMPU® bracelet.

A standardized questionnaire will be administered to each mother to collect information on socio-demographic characteristics and contact information. As is the standard of care, all mothers regardless of study arm will be taught how to provide KMC, how to monitor the infant's condition and recognize dangerous clinical signs during KMC and will be supported by a nurse during initial attempts at practicing KMC.

Mothers of infants randomly allocated to the intervention arm will be taught to use the bracelet. The meaning of the audiovisual alarm will be explained as well as the measures to be taken if the device indicates any sign of hypothermia. There will not be any additional training beyond that pertaining to the BEMPU® bracelet. The study nurse will then place the BEMPU® bracelet on the wrist of the infant. Infants in the intervention arm will wear the bracelet for up to 28 days post-discharge.

After discharge, participants in both the intervention and control arms will receive two study visits; one at 7 days post discharge and one at 28 days post-discharge. During each visit, infants will receive a physical examination to collect weight, length, head circumference and axillary temperature, and additional data will be collected on history of illnesses, care-seeking and treatment, KMC and feeding practices, and frequency of use of the bracelet (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Currently being treated in the KMC or neonatal ward at one of the participating hospitals
* Age<28 days
* Weight <2,500 grams at birth
* Clinically stable
* Mother is available, willing and able to provide consent

Exclusion Criteria:

* Clinically unstable
* Twin or multiple birth
* Ineligible to initiate KMC
* Mother <18 years of age
* Residence outside health facility catchment area or intention to relocate during the four weeks following discharge

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 380 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Hypothermia | up to 28 days
  Axilliary temperature <36.5 degrees Celsius assessed at 7 days

SECONDARY OUTCOMES:
Weight gain | 7 days and 28 days
  Change in weight in grams assessed at 7 days and 28 days
Kangaroo Mother Care | 7 days and 28 days
  Proportion of babies who received KMC for at least 8 hours in the last 24 hours assessed at 7 days and 28 days
All cause mortality | 28 days
  Number of neonatal deaths
Exclusive breastfeeding | 7 days and 28 days
  Proportion of babies who were exclusively breastfed in the last 24 hours assessed at 7 days and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mufaro Kanyangarara, Principal Investigator — University of South Carolina; Prince Owusu, Principal Investigator — Centre for Learning and Childhood Development - Ghana
Locations (6):
- Ghana (6):
  - Achimota General Hospital, Accra
  - Greater Accra Regional Hospital, Accra
  - Korle-Bu Teaching Hospital, Accra
  - Princess Marie Luis Children's Hospital, Accra
  - Central Regional Hospital, Cape Coast
  - Eastern Regional Hospital, Koforidua

IPD SHARING:
Plan to Share IPD: No